CLINICAL TRIAL: NCT05981677
Title: Risk and Social Feedback in Adolescents With Nonsuicidal Self-Injury
Brief Title: Social Feedback and Dysfunctional Risk Taking in NSSI Adolescents
Status: Recruiting | Type: Observational
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Benjamin Becker, Professor, University of Electronic Science and Technology of China
Other Study IDs: BAM_lab_NSSI_03
Record Dates: First submitted 2023-07-20; First posted 2023-08-08 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Nonsuicidal Self Injury; Risk-Taking
MeSH Terms: conditions — Self-Injurious Behavior; Risk-Taking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NSSI
- HC

SUMMARY:
Nonsuicidal self-injury (NSSI) is defined as direct, intentional physical injury without suicidal intention. Problematic interpersonal relationships and decision-making have been demonstrated to play crucial roles in this maladaptive behavior, especially for adolescents. Accumulating evidence suggests that decision processes and risk-taking are strongly influenced by the affective state of the individual. However, whether these interactions are disrupted in NSSI adolescents has not been systematically examined. In the current study, the investigators modified one of the most widely used paradigms for measuring an individual's risk decision-making, the Balloon Analogue Risk Task (BART). The investigators combine social reward (green balloon), punishment (red balloon), and control feedback (yellow balloon), to investigate whether the NSSI adolescents have dysfunctional risk-taking behavior while facing different social outcomes. The investigators recruit one group of NSSI adolescents (n = 40) and one health control (HC) group (n = 40), to compare their risk-related decisions during the emotional BART. The investigators hypothesize that compared to HC, NSSI adolescents will show altered effects of social reward and punishment on risk-related decision-making, in particular higher risk avoidance in the context of social punishment.

ELIGIBILITY:
Inclusion Criteria:

* 15-18 years
* right-handed
* normal or corrected normal visual acuity
* meet the proposed DSM-5 frequency criteria (e.g., ≥5 days of NSSI behaviors in the past year)

Exclusion Criteria:

* diagnosis of borderline personality disorder, major depressive disorder, other
* psychiatric disorders, etc.
* high suicidal risk
* recent use of medications that can affect neural activity
* have received or are receiving Dialectical Behavior Therapy (DBT) other treatment for emotional problems within the past 6 months
* have a contraindication to MRI scanning (e.g., metal implants, claustrophobia or other conditions that make them inappropriate for MRI scanning)

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Treatment-seeking NSSI individuals will be recruited from local hospitals and HC from the community.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Risky avoidance measured by BART | About 20 minutes
  Adjusted number of pumps (average number of pumps excluding balloons that exploded) as the index of risk avoidance. Alterations in the patients will be determined by using ANOVA models with the group (NSSI vs. HC) as a between-subject factor and emotional feedback (social reward, social punishment, and control) as a within-subject factor.
Decision-making measured by BART | About 20 minutes
  Earned money (total amount of money earned in the task) as the index of decision-making. Alterations in the patients will be determined by using ANOVA models with the group (NSSI vs. HC) as a between-subject factor and emotional feedback (social reward, social punishment, and control) as a within-subject factor.

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Provincial Center for Mental Health, Sichuan Provincial People's Hospital, University of Electronic Science and Technology of China, Chengdu, Sichuan, China